CLINICAL TRIAL: NCT03010995
Title: The Acute Cardiovascular Effects of Nicotine in E-cigarettes (ACE) Study
Acronym: ACE
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study discontinued due to lack of study funding.
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Affan B. Irfan, Principal investigator, University of Louisville
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 16.1079
Record Dates: First submitted 2016-12-09; First posted 2017-01-05 (Estimated); Last update posted 2018-07-26 (Actual); Status verified 2018-07

CONDITIONS: Cigarette Smoking Toxicity; Nicotine; Acute Cardiovascular Disease
Keywords: electronic cigarette; endothelial function
MeSH Terms: conditions — Vaping | interventions — Prazosin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All the outcome measurements will be performed by staff that will be blinded to the participant and their exposure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 18 mg nicotine (Active Comparator): E-cigarette with 18 mg nicotine
  Interventions: Drug: Prazosin
- 9 mg nicotine (Active Comparator): E-cigarette with 9 mg nicotine
  Interventions: Drug: Prazosin
- 0 mg nicotine (Placebo Comparator): E-cigarette with 0 mg nicotine
  Interventions: Drug: Prazosin

INTERVENTIONS:
Drug: Prazosin — Prazosin will used to study the mechanism involved in nicotine induced acute cardiovascular changes

SUMMARY:
The goal of this project is to evaluate the nicotine induced acute cardiovascular changes in E-Cigarette users and also study the mechanism involved particularly with vascular impairment.

DETAILED DESCRIPTION:
We will recruit 30 experienced E-cigarette users (those using E-Cigarette for at least 1 month and ≤ 1 tobacco cigarette / day), between ages 21-40 years; in 4 day study visit and 10 non-smokers (those who used less than 100 tobacco cigarettes in their lifetime and not active nicotine/tobacco or related product user) for a one study visit.The participants will be asked to abstain from all tobacco/nicotine and related product use for 12 hours before each visit.

Measurements will be taken at each study visit before and after E-cigarette use, each day with different nicotine dose, to look at both the individuals' exposure to nicotine and also the effects on the cardiovascular system. These measurements will include blood and urine samples as well as non-invasive cardiovascular measurements.

ELIGIBILITY:
Inclusion Criteria:

1. Participant will be currently healthy individuals, between 18 and 40 years of age.
2. E-Cigarette users using E-Cigarette for at least 1 month and smoke ≤ 1 tobacco cigarette / day; non-smokers who used less than 100 tobacco cigarettes in their lifetime and are not active nicotine/tobacco or related product users
3. Participants willing to abstain from vaping, smoking and tobacco for 12 hours prior to study.
4. Do not meet any of the Exclusion criteria.

Exclusion Criteria:

1. Unwilling or unable to provide informed consent.
2. Participant that have: Diabetes, Hypertension HIV, hepatitis, liver disease (including fatty liver), anemia, unhealed wounds, active infection, febrile, anemia, organ transplant, renal replacement therapy, kidney disease or insufficiency, dialysis, active cancer of any type, and untreated thyroid disease, major injury or trauma.
3. Body weight less than 100 pounds or BMI >40.
4. Participants that are taking the following medications: estrogen, testosterone, anti TNF agents, cyclophosphamide, ketoconazole, methoxsalen, pilocarpine, Isoniazid, rifampicin certain biologics, or Procrit
5. Participants that are currently using nicotine patches, nicotine gum or any form of nicotine-containing cessation device
6. Pregnant or lactating women.
7. Prisoners and other vulnerable populations.
8. Anyone that PI thinks is unsafe to participate in the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Change between baseline and post exposure 20-30 mins
  Flow mediated dilatation

SECONDARY OUTCOMES:
Heart rate | Change between baseline and post exposure 5,10, 30, 60, 120 mins
  Heart rate monitor
Blood pressure | Change between baseline and post exposure 5,10, 30, 60, 120 mins
  Blood pressure monitor
Heart Rate Variability | Change between baseline and post exposure 20 mins
  SphygmoCor HRV system SCOR-Hx
Nicotine levels in plasma | Change between Baseline and over 2 hours
  Detect plasma nicotine levels

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No